CLINICAL TRIAL: NCT04579315
Title: Long-term Effects of the New Nordic Renal Diet on Phosphorus and Lipid Homeostasis in Patients With Chronic Kidney Disease, Stages 3 and 4 - A Randomized Controlled Trial
Brief Title: Long-term Effects of the New Nordic Renal Diet in Patients With Moderate Chronic Kidney Disease
Acronym: CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bo Feldt-Rasmussen (Other)
Responsible Party: Sponsor-Investigator, Bo Feldt-Rasmussen, Professor, MD, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-20026376
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Chronic Kidney Disease(CKD); Hyperphosphatemia; Blood Pressure
Keywords: Chronic kidney disease; CKD; Phosphorus; Nutritional intervention; New Nordic Diet
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia

STUDY DESIGN:
Intervention Model Description: Two arms, one intervention group and one control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group, NNRD group (Active Comparator): Main principles of the interventional whole food approach are:
  * Maximum of 850 mg phosphorous/day
  * Protein: 0.8 g/kg/day
  * 80% vegetable products; 20% animal products
  * Maximum of 5-7 g NaCl/day (table salt)
  * Fresh raw products
  * Seasonal oriented
  * Fish: At least once a week
  * Vegetarian: At least once a week
  * Wide range of fruit and vegetables
  * Easy to follow in daily practice
  * Rich in flavors
  * Sufficient content of micro- and macronutrients
  Interventions: Other: Intervention group; NNRD group
- Control group (No Intervention): There is no intervention, patients are following their habitual diet

INTERVENTIONS:
Other: Intervention group; NNRD group — The intervention is a whole food approach, meaning that the participants in the intervention group receives all daily food elements that they should consume
  Arms: Intervention group, NNRD group

SUMMARY:
As Chronic Kidney Disease (CKD) progresses normophosphatemia is maintained by increasing the per nephron urinary phosphorus excretion. Clinically, hyperphosphatemia is associated with high mortality, vascular calcification, endothelial dysfunction and progression of left ventricular hypertrophy. Currently the treatment of hyperphosphatemia is first being initiated in stage 5 and consists of dietetic guidance to avoid dietary phosphate and treatment with oral phosphate binders. However, studies have shown important side effects to phosphate binders in terms of progression of vascular calcifications. Therefore, it might be beneficial to start the dietetic treatment with a reduction of dietary phosphate earlier in the disease stage.

The aim of this project is to develop a New Nordic Renal Diet (NNRD) for CKD patients' stage 3-4 and to examine the long-term effects in a period of 26-weeks. NNRD has a high content of vegetable foods, less animal products and more local food items with a lesser content of phosphorus.

DETAILED DESCRIPTION:
This study is a randomized controlled trial performed at Department of Nephrology Rigshospitalet, Copenhagen Denmark. Sixty patients will be randomized to either 26 weeks on the NNRD (intervention) or 26 weeks on their habitual diet (control). The patients will be randomized by blinded drawing by lot. The study participants can leave the trial at any time during the study period, without any explanation. The investigator can at any time pull a patient out of the trial, if there is concern for the patient's safety or if there is a breach in terms of following the protocol. The principal investigator is required to document and report dropouts from the study.

The project group has entered a cooperation agreement with Danish chefs. The agreement involves that a team consisting of highly talented chefs will create the recipes for the intervention. The recipes will be created in close collaboration with the principal investigator who will use her expertise within Clinical Nutrition to combine the international nutrients guidelines and culinarian experiences. Moreover, the agreement holds that they will find the raw materials needed for the recipes and deliver them weekly to the patients' homes throughout the study period in packages containing the recipes and raw materials. There will be no financial costs for the patients. The patients in the intervention group are expected to follow the recipes five days of the week during the study period. The final two days of the week, the patients must plan their own meals. However, still following the recommended guidelines upon the NNRD whole food approach delivered from the principal investigator, who is a phd.-student and also a registered clinical dietitian and MSc in clinical nutrition (Nikita Misella Hansen).

Sample size calculation and statistical analysis:

The sample size calculation is based on results from previous studies performed by this study group. Within 6 months of participating in this study we expect a decrease in eGFR to be about 1 ml/min/1.73 m2. This will have no influence on the total amount of 24-h urine phosphorus excretion (primary endpoint), as CKD progresses normophosphatemia is maintained by increasing the per nephron urinary phosphorus excretion stimulated by an increase in FGF23 and PTH leading to progressively increasing plasma levels of FGF23 and SHP the "phospho-toxicity model hypothesis" to a compensation from PTH and FGF23. In a randomized controlled study with a type-1-error risk of 0.05 (alfa, two tailed) and a power of 80% (beta) with a standard deviation of 24-h urine phosphorus excretion of 200 mg and a minimum clinical relevant difference of 300 mg the study population is estimated to 21 in each group. In case of drop-outs we will include 30 participants in each group. Therefore, total number of patients to be included in this study is 60.

Timeline for the study:

1. Baseline (day 0)

   Written consent will be obtained, randomization will be performed, and the following data will be registered:
   * Patient history: Gender, age, disease history, current medical record, diagnoses
   * Comorbidities - e.g. cardiovascular diseases, chronic obstructive lung disease, diabetes, hyperlipidemia, hypertension
   * Smoking (years) and alcohol consumption (average per week)
   * Blood- and urine samples
   * DEXA-scan and Electrocardiogram (ECG)
   * Blood pressure
   * Weight, BMI, hip- and waist circumference
   * Questionnaires regarding quality of life
   * Dietary record
2. Day 14 The patients will be asked to deliver a 24-hour urine sample for measuring phosphorus excretion. Furthermore, blood samples will be drawn
3. Day 30, 60, 90, 120, 150

   Every 4th week during the study period of 26 weeks (a total of 6 times) all patients will be evaluated at the Department of Nephrology, University Hospital, Copenhagen. During these first 5 visits the following data will be gathered:
   * 24-h urine phosphorus excretion
   * Blood samples
   * Blood pressure
   * Weight, hip- and waist circumference
4. Once a week Once every week the principal investigator will offer all the patients a telephone meeting. Duration of the phone conversation will depend on individual needs, but up to 20 minutes per patient/week despite of allocation. The content of these conversations will evolve around dietary intake and overall general condition. The principal investigator is in close collaboration with the others in the research group who are all medical doctors and will discuss any clinical problem if needed.
5. Day 180 (study completion)

   During the last day of the study period, the patients will be asked to meet at Rigshospitalet one more time. Data as on day 30, 60, 90, 120 and 150 will be gathered, moreover the following information will be obtained:
   * DEXA-scan and ECG
   * Weight, BMI, hip- and waist circumference
   * Questionnaires regarding quality of life
   * Dietary record
6. Follow-up visit Three months after study completion there will be an end-of-trial visit with a 24-h urine collection and blood samples

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Estimated glomerular filtration rate (eGFR) 20-45 ml/min
* Medically stable for two months prior to study start
* Written and verbally information is given
* Read, speak and understands Danish
* Written consent

Exclusion Criteria:

* Treatment with phosphate binders
* Metabolic disorders that requires specific dietary regulation
* Treatment with chemotherapy within the past 6 months
* Pregnancy and breastfeeding
* Food allergies
* Vegans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Difference in change in 24-hour urine phosphorus excretion from baseline to week 26 between the two study groups | Baseline, day: 14, 30, 60, 90, 120, 150, 180 and three months after study completion
  24-hour urine sample

SECONDARY OUTCOMES:
Difference in changes from baseline to week 26 between study groups in urinary excretion of calcium - creatinine, -urea and protein | Baseline, day: 14, 30, 60, 90, 120, 150, 180 and three months after study completion
  24-hour urine sample
Difference in changes from baseline to week 26 between study groups in blood lipids | Baseline, day: 14, 30, 60, 90, 120, 150, 180 and three months after study completion
  Blood samples
Difference in changes from baseline to week 26 between study groups in FGF23, Fractional excretion of phosphorus, P-phosphate, P-calcium, P-PTH, P-1,25OH2vitamin D3 and P-albumin | Baseline, day: 14, 30, 60, 90, 120, 150, 180 and three months after study completion
  Blood samples
Difference in changes from baseline to week 26 between study groups in glomerular filtration rate, as judged by P-creatinine | Baseline, day: 14, 30, 60, 90, 120, 150, 180 and three months after study completion
  Blood samples
Difference in changes from baseline to week 26 between study groups in weight | Baseline, day: 30, 60, 90, 120, 150, 180 and three months after study completion
  Weight changes in kilograms
Difference in changes from baseline to week 26 between study groups in hip- and waist circumferences | Baseline, day: 30, 60, 90, 120, 150, 180 and three months after study completion
  Hip/waist circumferences in centimeters
Difference in changes from baseline to week 26 between study groups in bone mineral density using DEXA scan (Dual-energy X-ray absorptiometry) | Baseline and study completion (day 180)
  Body composition, focusing on bone mineral density using DEXA scan (Dual-energy X-ray absorptiometry)
Difference in changes from baseline to week 26 between study groups in blood pressure, both systolic and diastolic blood pressure | Baseline, day: 30, 60, 90, 120, 150, 180 and three months after study completion
  Blood pressure mm Hg (systolic and diastolic)
Difference in changes from baseline to week 26 between study groups in quality of life | Baseline and study completion (day 180)
  Scale EQ-5D-5L questionnaire. Low/high scores varies in terms of reflecting better or worse outcomes
Dietary satisfaction in the intervention group | Day 30, 60, 90, 120, 150, 180
  5-likert scale questionnaire. Low/high scores varies in terms of reflecting better or worse outcomes
Difference in changes from baseline to week 26 between study groups in SuPAR and GDF15 | Baseline, day: 14, 30, 60, 90, 120, 150, 180 and three months after study completion
  Blood samples
Difference in change in metabolic acidosis from baseline to week 26 between the two study groups | Baseline, day: 14, 30, 60, 90, 120, 150, 180 and three months after study completion
  24-hour urine sample

CONTACTS AND LOCATIONS:
Overall Officials: Bo Feldt-Rasmussen, Professor, Study Chair — Department of Nephrology, Rigshospitalet, Copenhagen Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
There is no current plan to make IPD available

REFERENCES:
- [Derived] Misella Hansen N, Kamper AL, Rix M, Feldt-Rasmussen B, Leipziger J, Sorensen MV, Berg P, Astrup A, Salomo L. Health effects of the New Nordic Renal Diet in patients with stage 3 and 4 chronic kidney disease, compared with habitual diet: a randomized trial. Am J Clin Nutr. 2023 Nov;118(5):1042-1054. doi: 10.1016/j.ajcnut.2023.08.008. Epub 2023 Aug 19. PMID 37598748
- [Derived] Hansen NM, Rix M, Kamper AL, Feldt-Rasmussen B, Christoffersen C, Astrup A, Salomo L. Study protocol: long-term effect of the New Nordic Renal Diet on phosphorus and lipid homeostasis in patients with chronic kidney disease, stages 3 and 4: a randomised controlled trial. BMJ Open. 2021 Aug 30;11(8):e045754. doi: 10.1136/bmjopen-2020-045754. PMID 34462278